CLINICAL TRIAL: NCT06296940
Title: Project WEST (Written Exposure in Substance Treatment) Part 2
Brief Title: Written Exposure in Substance Treatment
Acronym: WEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Potomac Health Foundations (Other)
Collaborators: University of Maryland, Baltimore County (Other)
Responsible Party: Principal Investigator, Rebecca Schacht, Affiliated Research Scientist, Potomac Health Foundations
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WEST 2.0
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-03

CONDITIONS: Posttraumatic Stress Disorder; Substance Use Disorders
Keywords: Written Exposure Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: We are conducting a randomized controlled trial of approximately 50 randomized subjects (up to 100 total enrollments) who will be assigned 1:1 to treatment as usual (TAU) or TAU+WET.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment as Usual (TAU) (Active Comparator): Participants randomized to the TAU condition, which involves the standard clinical services available in a short term residential SUD treatment context. Examples of these services are: Individual counseling/case management; Group psychoeducation; Group counseling; Assessment and addiction related medical treatment from a physician; Pharmacotherapy for substance use disorders; 12-step groups. However, participants in this group do not receive treatment that is targeted at decreasing PTSD symptoms.
  Interventions: Behavioral: Treatment as Usual
- TAU + Written Exposure Therapy (WET) (Experimental): Participants in this condition receive everything included in TAU plus 5 individual sessions of WET delivered by a therapist. Sessions average less than 60 minutes and primarily involve writing about the traumatic experience that is guided by the therapist.
  Interventions: Behavioral: Written Exposure Therapy; Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Written Exposure Therapy — Written Exposure Therapy is a brief, evidenced based intervention for PTSD. WET is generally delivered individually across 5 sessions in which the therapist guides the patient through writing exercises. Across exposure sessions, participants experience habituation so that their symptoms decrease by the end of treatment. WET has an established evidence base in general outpatient psychotherapy for PTSD, but has not been adapted or tested in residential SUD treatment settings.
  Arms: TAU + Written Exposure Therapy (WET)
Behavioral: Treatment as Usual — Treatment as Usual will include a variety of standard care services offered in short term residential treatment. For example, participants receiving TAU will participate in individual case management/general counseling sessions focused on their substance use disorder and its consequences, group based psychoeducation sessions, group based counseling sessions (e.g., relapse prevention planning), individual services with a medical provider and pharmacotherapy (e.g., for withdrawal, relapse prevention, or co-occurring conditions)

SUMMARY:
The purpose of this pilot randomized clinical trial is to test the feasibility and efficacy of written exposure therapy (WET) for posttraumatic stress disorder (PTSD) within the context of residential substance use disorder (SUD) treatment. All participants meet criteria for PTSD and are in a short term residential SUD treatment program (target residential treatment duration = 28 days) regardless of the research. The main questions the study aims to answer are: 1) Is the delivery of WET feasible in short term residential SUD treatment for individuals with severe SUD; 2) Do participants in the TAU+WET condition have greater reductions in PTSD symptoms pre/post treatment compared to participants in TAU alone?

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Fluent in English
* Cognitively able to provide consent to the research
* Enrolled in inpatient treatment at the clinical site where the research takes place
* Meet criteria for probable PTSD based on PCL-5 score
* Be early enough in their residential stay to allow time to complete the WET protocol
* Have a clear memory of the traumatic event so they are able to write about itin detail

Exclusion Criteria:

* Reports significant suicidal or homicidal ideation with intent, untreated psychosis, or have other health limitations that may interfere with their ability to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of WET | Pre/post intervention window (approximately 3 weeks)
  PTSD symptom reduction pre/post intervention by treatment arm as measured by the posttraumatic checklist for DSM-5 (PCL-5). The PCL-5 is a self-report questionnaire yielding scores ranging from 0-80 with higher scores indicating greater symptomology.

SECONDARY OUTCOMES:
Feasibility of WET delivered in residential SUD treatment context | Up to 4 weeks, or until the participant discharges from residential treatment (whichever comes first).
  Percentage of participants in the WET arm who were able to complete the treatment (5 sessions) prior to discharge
Acceptability of WET delivered in residential SUD treatment context | Collected post intervention window (approximately 3 weeks from randomization)
  Treatment satisfaction scores among WET participants as measured by the 2-part credibility/expectancies questionnaire (CEQ). The CEQ utilizes two scoring systems that range from 1-9 or 0%-100%. with higher scores indicating greater acceptability.

CONTACTS AND LOCATIONS:
Locations (1):
- Maryland Treatment Centers, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD may be shared with other researchers through a de-identified, secure, electronic data transfer as allowed by the IRB and other regulatory authorities.
Time Frame: Interested individuals may inquire after data lock is achieved and the primary outcomes paper has been published from this dataset. Estimated time: 2026

REFERENCES:
- [Background] Schacht RL, Wenzel KR, Meyer LE, Mette M, Mallik-Kane K, Rabalais A, Berg SK, Fishman M. A pilot test of Written Exposure Therapy for PTSD in residential substance use treatment. Am J Addict. 2023 Sep;32(5):488-496. doi: 10.1111/ajad.13442. Epub 2023 Jun 17. PMID 37329251